CLINICAL TRIAL: NCT04045132
Title: Social Media-Based Parenting Program for Women With Postpartum Depressive Symptoms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Philadelphia (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 19-016174; R61MH118405 (NIH); 19-016174-B (Other: Children's Hospital of Philadelphia)
Record Dates: First submitted 2019-08-01; First posted 2019-08-05 (Actual); Results first posted 2022-02-11 (Actual); Last update posted 2023-12-27 (Actual); Status verified 2023-12

CONDITIONS: Postpartum Depression; Parenting; Parent-Child Relations
Keywords: Social Media; Postpartum Depression; Parenting; Infants; Mothers
MeSH Terms: conditions — Depression, Postpartum

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Video coders will be blinded to intervention assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MoodGym Alone (Active Comparator): The MoodGym program is an evidence-based online cognitive behavioral treatment program that has been shown to be effective at reducing depression symptoms in a meta-analysis of 11 trials (g=0.36, 95% CI 0.17-0.56). Moodgym contains five modules with interactive exercises, workbooks, anxiety and depression quizzes, and downloadable relaxation audio files that can be completed online without therapist interaction.
  Interventions: Behavioral: MoodGym
- Parenting Program + MoodGym (Experimental): The social media-based parenting program consists of 8 weekly sessions using a Facebook platform with the following topics: depression psychoeducation and behavioral activation, infant temperament, play, feeding, safety, sleep, parent-child interactions, and shared book reading. Participants in the experimental arm will also be enrolled in the online depression treatment program, MoodGym.
  Interventions: Behavioral: Social Media-Based Parenting Program; Behavioral: MoodGym

INTERVENTIONS:
Behavioral: Social Media-Based Parenting Program — Participants in the intervention group will be enrolled in Facebook secret user groups, administered by a trained facilitator, in order to permit participants to view and comment on posted materials. Content and user identity are restricted to invited participants to maintain privacy. For each topic, we organize educational materials into video vignettes, narrated PowerPoint presentations, and written materials. The facilitator reviews and comments on postings daily, provides feedback to participants, and removes inappropriate postings if they occur. Facebook analytics for the secret groups are available to group administrators and will provide information on any sessions viewed (engagement) and counts of sessions viewed and comments posted (dosage). Women in the intervention group will also be enrolled in the online depression treatment program, MoodGym.
  Arms: Parenting Program + MoodGym
Behavioral: MoodGym — Participants in the control group will be enrolled in MoodGym, an evidence-based online Cognitive Behavioral Therapy (CBT) program for depression. Through the MoodGym program, participants will have access to interactive exercises, workbooks, anxiety and depression quizzes, and downloadable relaxation audio files. We will supplement Moodgym with a facilitator contact by texting or email to check-in and encourage completion of intervention. MoodGym will provide information on the number of sessions completed by participants (engagement and dosage).

SUMMARY:
The purpose of this study is to determine whether a social media-based parenting program can improve responsive parenting among mothers with Postpartum depression (PPD) symptoms. Participants will be randomized to receive the parenting program plus online depression treatment or online depression treatment alone to assess target engagement. Our overall objective for this application is to study whether this program combined with online depression treatment leads to more responsive parenting (target) and signals improved child language, socioemotional and cognitive development (outcomes) compared to depression treatment alone.

DETAILED DESCRIPTION:
Postpartum depression (PPD) symptoms are common among women following the birth of a child and can adversely impact a mother's ability to care for her child. As a result, infants of mothers with PPD symptoms may experience less responsive parenting, placing them at greater risk for delays in development. Evidence- based parenting programs have been developed to guide mothers with caring for their infants but may not address the impact of depression on parenting, are intensive and expensive to administer with limited ability for scale up, or are not available in a format that facilitates participation by women with depressive symptoms. To address these barriers, we developed a theoretically-driven social media-based parenting program on responsive parenting and child development.

To determine whether the social media-based parenting program can improve responsive parenting among women with PPD symptoms, we will conduct a prospective individually randomized group treatment trial. 75 eligible women who screen positive for PPD at their infants' well child visit and their children will be consented, enrolled, and randomized as mother-child dyads 1:1 to receive a) the social media-based parenting program plus online depression treatment or b) online depression treatment alone. We chose a randomized design, because it is most effective in guarding against bias and will ensure that patients in both arms are similar in observed and unobserved characteristics. Treatment assignment will be done at the time of enrollment following informed consent.

Descriptive statistics for demographic and poverty characteristics and PPD symptoms measured at baseline will be examined across the two treatment groups to assess the success of the randomization. We will assess responsive parenting at baseline and 3 months post-enrollment. Secondary outcomes, including changes in EPDS, BDI-II PSOC, and PSI-SF scores measured between baseline and the 3-month follow-up between groups, will be explored to determine if the effects of the parenting program are consistent with preliminary pilot findings. The intervention arm will also be assessed with the Therapeutic Factors Inventory-8 (TFI-8) to measure cohesion and the Acceptability survey which measures feasibility of the parenting program at 3-months post-enrollment. Additionally, at the 3-month mark, all participants will be administered the MoodGym Acceptability Survey to assess feasibility of the online depression treatment program.

The results of this application would be expected to contribute important new knowledge and inform a future trial on parenting strategies to better assist mothers with PPD symptoms and improve child developmental outcomes.

ELIGIBILITY:
Inclusion Criteria:

Women who:

* Are >18 years old
* Screen positive for postpartum depression (score>9) on the EPDS at a participating pediatric practice
* Have an infant <8 months of age
* Speak and Read English
* Have Access to a smart phone or computer tablet with internet access

Children who:

* Are < 8 months old

Exclusion Criteria:

Women who:

* Report suicidality (i.e., suicidal ideation and/or behavior) on the EPDS (Question #10) at enrollment.
* Report severe depressive symptoms (EPDS>20) at enrollment.
* Have a substantiated report of child maltreatment

Children who:

* Were born premature (estimated gestational age<35 weeks)
* Have been diagnosed with congenital malformations or genetic syndromes which place them at risk of developmental delays
* Are already currently receiving early intervention services for developmental delays at baseline

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2019-12-17 (Actual); Primary Completion 2021-10-07 (Actual); Study Completion 2021-10-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James Guevara, MD, MPH, Principal Investigator — Children's Hospital of Philadelphia; Rhonda Boyd, PhD, Principal Investigator — Children's Hospital of Philadelphia
Locations (1):
- Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
A complete, cleaned, and de-identified dataset will be made available to other investigators after all analyses have been conducted and within twelve months of the end of the final year of funding to allow for publication of all study aims. To obtain this data set, other investigators will need to contact the study Principal Investigator (PI) who will provide a data sharing agreement. The data sharing agreement will permit a deidentified data set to be shared once an Institutional Review Board (IRB) protocol has been approved at the investigators' home institution and the investigators have signed a pledge to not attempt to identify individual study subjects. The data set will be made available on a Compact Disc Read-Only Memory (CD-ROM) or through a secure File Transfer Protocol (FTP) site.
Supporting Information: Study Protocol, SAP
Time Frame: 12 months after the end of the final year of funding.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: From December 2019 to March 2020, recruitment took place over the phone and enrollment was completed on site at the Roberts Center for Pediatric Research at the Children's Hospital of Philadelphia. Due to the COVID-19 pandemic, there was a recruitment pause from March-June 2020. As of June 12th, 2020, the study was approved by the IRB to enroll participants to the study virtually, and remaining recruitment and enrollment activities were completed virtually.
Pre-assignment Details: If a participant was enrolled to the study but did not complete the videotaped baseline Parent Child Early Relational Assessment before the start of the intervention, regardless of the group they were randomized to, they were withdrawn from the study.
Groups:
- MoodGym Alone (Control): The MoodGym program is an evidence-based online cognitive behavioral treatment program that has been shown to be effective at reducing depression symptoms in a meta-analysis of 11 trials (g=0.36, 95% CI 0.17-0.56). Moodgym contains five modules with interactive exercises, workbooks, anxiety and depression quizzes, and downloadable relaxation audio files that can be completed online without therapist interaction.
  MoodGym: Participants in the control group will be enrolled in MoodGym, an evidence-based online Cognitive Behavioral Therapy (CBT) program for depression. Through the MoodGym program, participants will have access to interactive exercises, workbooks, anxiety and depression quizzes, and downloadable relaxation audio files. We will supplement Moodgym with a facilitator contact by texting or email to check-in and encourage completion of intervention. MoodGym will provide information on the number of sessions completed by participants (engagement and dosage).
- Parenting Program + MoodGym (Intervention): The social media-based parenting program consists of 8 weekly sessions with the following topics: depression psychoeducation and behavioral activation, infant temperament, play, feeding, safety, sleep, parent-child interactions, and shared book reading. Participants in the experimental arm will also be enrolled in the online depression treatment program, MoodGym.
  Social Media-Based Parenting Program: Participants in the intervention group will be enrolled in Facebook secret user groups. Content and user identity are restricted to invited participants to maintain privacy. For each topic, we organize educational materials into video vignettes and written materials. The facilitator reviews and comments on postings daily, provides feedback to participants, and removes inappropriate postings if they occur. Facebook analytics for the secret groups are available to group administrators and will provide information on any sessions viewed (engagement) and counts of sessions viewed and comments posted (dosage).
  MoodGym: Participants in the control and intervention groups will be enrolled in MoodGym, an evidence-based online Cognitive Behavioral Therapy (CBT) program for depression. Through the MoodGym program, participants will have access to interactive exercises, workbooks, anxiety and depression quizzes, and downloadable relaxation audio files. We will supplement Moodgym with a facilitator contact by texting or email to check-in and encourage completion of intervention.
Period: Overall Study
Arm/Group | MoodGym Alone (Control) | Parenting Program + MoodGym (Intervention)
Started (These numbers represent the participants who completed a baseline visit and were randomized.) | 37 | 38
Completed (These numbers represent the participants who at the 3-month follow up completed all secondary measures as well as the Parent Child Early Relational Assessment (PCERA). Those who did not complete the PCERA and/or who did not complete all the follow up measures were not considered to have completed their study participation.) | 34 | 32
Not Completed | 3 | 6
Not completed — Lost to Follow-up | 3 | 6

BASELINE CHARACTERISTICS:
Population: Participants who completed a Baseline Demographics measure were included in the overall analysis. At Baseline, 75 (37 control and 38 intervention) total enrolled participants completed the Demographics measure.
Groups:
- Total: Total of all reporting groups
Arm/Group | MoodGym Alone (Control) | Parenting Program + MoodGym (Intervention) | Total
Number analyzed (Participants) | 37 | 38 | 75
Age, Continuous [Mean (Standard Deviation); unit: years] | 28.5 (4.8) | 29.8 (5.6) | 29.2 (5.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37 | 38 | 75
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 3
  Not Hispanic or Latino | 36 | 36 | 72
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: participants]
  American Indian/Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Black | 28 | 24 | 52
  >1 Race/Other | 1 | 3 | 4
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  White | 7 | 11 | 18
Region of Enrollment [Number; unit: participants]
  United States | 37 | 38 | 75
The Parent Child Early Relational Assessment (PCERA) [Mean (Standard Deviation); unit: score on a scale] — The Parent Child Early Relational Assessment is a 65-item videotape assessment designed to measure the quality of affect and behavior in parent-infant interactions. The PCERA has been shown to possess good interrater reliability, internal consistency, discriminant and concurrent validity, and sensitivity to change. 3 parenting subscales will be the focus. Each individual subscale is scored between 0-5, with higher scores indicating more responsive parenting. A subscale score of 1-2 indicates concern, a score of 3 indicates some concern, and a score of 4-5 of strength. Population: Participants who completed a Baseline Parent Child Early Relational Assessment (PCERA) videotape measure were included in the overall analysis. At Baseline, 73 (36 control and 37 intervention) of the 75 total enrolled participants completed a PCERA videotape measure. .
  score on a scale
    PCERA Factor 1 (Baseline)- Parental Positive Affective Involvement and Verbalization: number analyzed (Participants) | 36 | 37 | 73
    PCERA Factor 1 (Baseline)- Parental Positive Affective Involvement and Verbalization | 3.0 (0.6) | 3.2 (0.6) | 3.1 (0.6)
    PCERA Factor 2 (Baseline)- Parental Negative Affect and Behavior | 4.1 (0.7) | 4.0 (0.8) | 4.1 (0.8)
    PCERA Factor 3 (Baseline)- Parental Intrusiveness, Insensitivity, and Inconsistency | 3.1 (0.4) | 3.1 (0.7) | 3.1 (0.6)

OUTCOME MEASURES:

1. Primary Outcome: The Parent Child Early Relational Assessment (PCERA)
Description: The Parent Child Early Relational Assessment (PCERA) is a validated 65-item videotape assessment designed to measure the quality of affect and behavior in parent-infant interactions. The PCERA uses ratings that are based on observations of 5-minute videotaped interactions with parent-infant dyads engaged in free play. The PCERA has been shown to possess good interrater reliability, internal consistency, discriminant and concurrent validity, and sensitivity to change. The PCERA contains 8 subscales of which 3 parenting subscales will be the focus: 1) Parental Positive Affective Involvement and Verbalization, 2) Parental Negative Affect and Behavior, and 3) Parental Intrusiveness, Insensitivity, and Inconsistency. Each individual subscale is scored between 0-5, with higher scores indicating more responsive parenting. A subscale score of 1-2 indicates an area of concern, a score of 3 indicates some concern, and a score of 4-5 indicates an area of strength.
Time Frame: Baseline and 3 Months
Population: Participants who completed both a Baseline and 3-month follow-up Parent Child Early Relational Assessment (PCERA) videotape measure were included in the overall analysis. At Baseline, 73 (36 control and 37 intervention) of the 75 total enrolled participants completed a PCERA videotape measure, and 66 (34 control and 32 intervention) of the 75 total enrolled participants completed a PCERA videotape measure at 3-month follow-up.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MoodGym Alone (Control) | Parenting Program + MoodGym (Intervention)
Number analyzed (Participants) | 36 | 37
score on a scale
  PCERA Factor 1 (Baseline)- Parental Positive Affective Involvement and Verbalization | 3.0 (0.6) | 3.2 (0.6)
  PCERA Factor 1 (3-month follow-up)- Parental Positive Affective Involvement and Verbalization: number analyzed (Participants) | 34 | 32
  PCERA Factor 1 (3-month follow-up)- Parental Positive Affective Involvement and Verbalization | 3.3 (0.5) | 3.3 (0.6)
  PCERA Factor 2 (Baseline)- Parental Negative Affect and Behavior | 4.1 (0.7) | 4.0 (0.8)
  PCERA Factor 2 (3-month follow-up)- Parental Negative Affect and Behavior: number analyzed (Participants) | 34 | 32
  PCERA Factor 2 (3-month follow-up)- Parental Negative Affect and Behavior | 4.3 (0.6) | 4.2 (0.8)
  PCERA Factor 3 (Baseline)- Parental Intrusiveness, Insensitivity, and Inconsistency | 3.1 (0.4) | 3.1 (0.7)
  PCERA Factor 3 (3-month follow-up)- Parental Intrusiveness, Insensitivity, and Inconsistency: number analyzed (Participants) | 34 | 32
  PCERA Factor 3 (3-month follow-up)- Parental Intrusiveness, Insensitivity, and Inconsistency | 3.5 (0.5) | 3.4 (0.6)

2. Secondary Outcome: The Edinburgh Postnatal Depression Scale (EPDS)
Description: The Edinburgh Postnatal Depression Scale (EPDS) is a validated 10-item self-report measure of depressive symptoms with strong evidence for reliability, validity, and utility in varying populations. It has been used extensively in mental health research and provides cutpoints to determine the severity of depressive symptoms. It includes a question on suicidal thoughts and wishes (#10) that will be used to monitor for suicidality. The total score (range: 0-30) will be used with scores of 10 or higher representing minor or moderate depression and scores of 20 or greater representing severe depression.These outcomes will assess changes in EPDS from baseline to 3 months.
Time Frame: Baseline, 1-month, 2-month, 3-month
Population: Participants who completed the Edinburgh Postnatal Depression Scale (EPDS) measure at each time point were included in the analysis. Over the 3-month time frame there were several participants who were lost to follow-up and did not complete the subsequent EPDS measures. This is the reason for the drop in number of participants analyzed between groups over the 3-month period.
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | MoodGym Alone (Control) | Parenting Program + MoodGym (Intervention)
Number analyzed (Participants) | 37 | 37
score on a scale
  EPDS Baseline | 15.2 [7 to 25] | 14.3 [7 to 20]
  EPDS 1-month follow-up | 12.6 [4 to 23] | 9.7 [3 to 19]
  EPDS 2-month follow-up | 11.7 [5 to 28] | 9.7 [2 to 19]
  EPDS 3-month follow-up: number analyzed (Participants) | 36 | 34
  EPDS 3-month follow-up | 10.1 [0 to 19] | 9.0 [1 to 22]

3. Secondary Outcome: The Beck Depression Inventory (BDI-II)
Description: The Beck Depression Inventory (BDI-II) is a 21-item self-report tool that measures the severity of depression and includes two subscales: cognitive and somatic. It has been well validated, and widely used, with scores 14-19 indicating mild depression, 20-28 moderate depression, and 29-63 severe depression. The total score (range: 0-63) will be used, with higher scores indicating higher levels of depression. These outcomes will assess changes in BDI-II from baseline to 3 months.
Time Frame: Baseline and 3-months
Population: Participants who completed the Beck Depression Inventory (BDI-II) measure at each time point were included in the analysis. At baseline there was one participant, of the 75 total enrolled, who did not complete any baseline measures, including the BDI-II. Over the 3-month time frame there were several participants who were lost to follow-up and did not complete the BDI-II measure. This is the reason for the drop in number of participants analyzed between groups over the 3-month period.
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | MoodGym Alone (Control) | Parenting Program + MoodGym (Intervention)
Number analyzed (Participants) | 37 | 37
score on a scale
  BDI-II Baseline | 23.6 [13 to 46] | 22.4 [5 to 41]
  BDI-II 3-month follow-up: number analyzed (Participants) | 36 | 34
  BDI-II 3-month follow-up | 14.6 [0 to 42] | 14.3 [1 to 40]

4. Secondary Outcome: The Parenting Sense of Competence Scale (PSOC)
Description: The Parenting Sense of Competence Scale (PSOC) is a validated 17-item self-report measure of parenting self-esteem and competence and consists of two factors: satisfaction and efficacy. Response categories are on a 6-point likert-scale from strongly disagree to strongly agree. The total score (range: 17-102), which includes the sum of the two factors, will be used. A higher score indicates a higher parenting sense of competency. There are no average scores or 'cut-off's' for this tool. These outcomes will assess changes in PSOC from baseline to 3 months.
Time Frame: Baseline and 3 months
Population: Participants who completed the Parenting Sense of Competence Scale (PSOC) measure at each time point were included in the analysis. At baseline there was one participant, of the 75 total enrolled, who did not complete any baseline measures, including the PSOC. Over the 3-month time frame there were several participants who were lost to follow-up and did not complete the PSOC measure. This is the reason for the drop in number of participants analyzed between groups over the 3-month period.
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | MoodGym Alone (Control) | Parenting Program + MoodGym (Intervention)
Number analyzed (Participants) | 37 | 37
score on a scale
  PSOC Baseline | 63.2 [48 to 80] | 63.9 [40 to 87]
  PSOC 3-month follow-up: number analyzed (Participants) | 36 | 35
  PSOC 3-month follow-up | 71.3 [55 to 93] | 71.1 [51 to 88]

5. Secondary Outcome: The Parenting Stress Index-Short Form (PSI-SF)
Description: The Parenting Stress Index-Short Form (PSI-SF) is a validated 36-item scale that measures parenting stress. The PSI-SF is a direct derivative of the full-length test (PSI) and it has been shown to have excellent internal consistency and to be positively associated with maternal psychological distress. Scores on the PSI-SF correlate well with the full-length PSI. It yields a Total Stress score from three scales: Parental Distress, Parent-Child Dysfunctional Interaction, and Difficult Child. The total score (range: 36-180) will be used, with higher scores indicating higher levels of stress.These outcomes will assess changes in PSI-SF from baseline to 3 months.
Time Frame: Baseline and 3 months
Population: Participants who completed the Parenting Stress Index-Short Form (PSI-SF) measure at each time point were included in the analysis. At baseline there was one participant, of the 75 total enrolled, who did not complete any baseline measures, including the PSI-SF. Over the 3-month time frame there were several participants who were lost to follow-up and did not complete the PSI-SF measure. This is the reason for the drop in number of participants analyzed between groups over the 3-month period.
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | MoodGym Alone (Control) | Parenting Program + MoodGym (Intervention)
Number analyzed (Participants) | 37 | 37
score on a scale
  PSI-SF Baseline | 89.2 [58 to 134] | 85.4 [48 to 115]
  PSI-SF 3-month follow-up: number analyzed (Participants) | 36 | 35
  PSI-SF 3-month follow-up | 75.5 [36 to 130] | 73.6 [38 to 108]

6. Secondary Outcome: The National Comorbidity Survey (NCS)
Description: The National Comorbidity Survey (NCS) provides data on mental health treatment in the United States. We will include a question from the NCS on prior mental health services use in the past month: "In the past month, did you receive treatment for problems with your emotions or nerves, or your use of alcohol or drugs?" We will consider mental health service use to have occurred in the past month if a mother responds "Yes" to this question. The results indicate the number of participants from each group who received mental health services/treatment at each time point. Additionally, if a mother responds "Yes" to the initial NCS item, a follow-up question will be asked to determine the specific types of services that were accessed: "If yes, what type of treatment did you receive?"
Time Frame: 1-month, 2-month, 3-month
Population: Participants who completed the National Comorbidity Survey (NCS) measure at each time point were included in the analysis. Over the 3-month time frame there were several participants who were lost to follow-up and did not complete the NCSmeasure. This is the reason for the drop in number of participants analyzed between groups over the 3-month period.
Measure: Count of Participants; unit: Participants
Groups:
- Parenting Program + MoodGym: The social media-based parenting program consists of 8 weekly sessions with the following topics: depression psychoeducation and behavioral activation, infant temperament, play, feeding, safety, sleep, parent-child interactions, and shared book reading. Participants in the experimental arm will also be enrolled in the online depression treatment program, MoodGym.
  Social Media-Based Parenting Program: Participants in the intervention group will be enrolled in Facebook secret user groups. Content and user identity are restricted to invited participants to maintain privacy. For each topic, we organize educational materials into video vignettes and written materials. The facilitator reviews and comments on postings daily, provides feedback to participants, and removes inappropriate postings if they occur. Facebook analytics for the secret groups are available to group administrators and will provide information on any sessions viewed (engagement) and counts of sessions viewed and comments posted (dosage).
  MoodGym: Participants in the control and intervention groups will be enrolled in MoodGym, an evidence-based online Cognitive Behavioral Therapy (CBT) program for depression. Through the MoodGym program, participants will have access to interactive exercises, workbooks, anxiety and depression quizzes, and downloadable relaxation audio files. We will supplement Moodgym with a facilitator contact by texting or email to check-in and encourage completion of intervention.
Arm/Group | MoodGym Alone | Parenting Program + MoodGym
Number analyzed (Participants) | 37 | 37
Participants
  NCS 1-month follow-up | 10 | 7
  NCS 2-month follow-up | 12 | 8
  NCS 3-month follow-up: number analyzed (Participants) | 36 | 34
  NCS 3-month follow-up | 11 | 10

7. Secondary Outcome: Multi-dimensional Scale of Perceived Social Support (MSPSS)
Description: The Multi-dimensional Scale of Perceived Social Support (MSPSS) is a 12-item scale that assesses perceived social support from family, friends, and a significant other. Response categories are on a 7-point likert-scale from 1=very strongly disagree to 7=very strongly agree. The total score will be used (range: 12-84).
Time Frame: Baseline
Population: Participants who completed a Baseline Multi-dimensional Scale of Perceived Social Support (MSPSS) measure were included in the overall analysis. At Baseline, 74 (37 control and 37 intervention) of the 75 total enrolled participants completed the MSPSS measure.
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | MoodGym Alone | Parenting Program + MoodGym
Number analyzed (Participants) | 37 | 37
score on a scale | 52.9 [12 to 84] | 58.0 [18 to 84]

8. Secondary Outcome: Therapeutic Factors Inventory (TFI-8)
Description: The TFI-8 is a validated 8-item scale that is used to measure cohesion and is continuous process monitoring for therapy groups. Scores on the TFI-8 correlate well with the full TFI. The total score (range: 8-56) will be used, with higher scores indicating greater cohesion within the group. The TFI-8 will be administered at the 3-month visit to the intervention group, only.
Time Frame: 3 months
Population: Participants in the Parenting Program + MoodGym (Intervention arm), only. At the 3-month time point, there were several participants who had been lost to follow-up and did not complete the TFI-8 measure. This is the reason for the drop in number of participants.
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | MoodGym Alone | Parenting Program + MoodGym
Number analyzed (Participants) | 0 | 34
score on a scale |  | 40.5 [18 to 56]

9. Secondary Outcome: Acceptability Survey
Description: The Acceptability survey is a 10-item scaled with 3 additional open ended questions that will be used to assess feasibility of the parenting program. The total score (range: 9-45) will be used and the open ended questions will be qualitatively analyzed to help inform the acceptability scores. Higher scores on the acceptability survey indicate greater satisfaction and feasibility of the parenting program. The acceptability survey will be administered at the 3-month visit to the intervention, only.
Time Frame: 3 months
Population: Participants in the Parenting Program + MoodGym (Intervention arm), only. At the 3-month time point, there were several participants who had been lost to follow-up and did not complete the Acceptability Survey measure. This is the reason for the drop in number of participants.
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | MoodGym Alone | Parenting Program + MoodGym
Number analyzed (Participants) | 0 | 34
score on a scale |  | 34.8 [17 to 45]

10. Secondary Outcome: MoodGym Acceptability Survey
Description: The MoodGym Acceptability survey will be used to assess feasibility of the online depression treatment program, MoodGym. The survey includes two qualitative open-ended questions and an additional question that asks, "It is ___________ that I will use MoodGym compared to going to a health care provider for depression treatment." The response is a 5-point likert-scale from "Much More Likely" to "Much Less Likely". The open ended questions will be qualitatively analyzed to help inform the acceptability scores. The MoodGym Acceptability survey will be administered at the 3-month visit to both the intervention and control group.
Time Frame: 3 months
Population: Participants who completed a 3-month MoodGym Acceptability Survey measure were included in the overall analysis. At the 3-month time point, there were several participants who had been lost to follow-up and did not complete the MoodGym Acceptability Survey measure. This is the reason for the drop in number of participants.
Measure: Count of Participants; unit: Participants
Arm/Group | MoodGym Alone | Parenting Program + MoodGym
Number analyzed (Participants) | 32 | 31
Participants
  Much More Likely | 7 | 6
  More Likely | 9 | 6
  No Difference | 7 | 11
  Less Likely | 3 | 4
  Much Less Likely | 6 | 4

ADVERSE EVENTS:
Time Frame: Adverse event data collected over the span of the 2-year study period
Description: The Children's Hospital of Philadelphia Institutional Review Board (IRB) defines a Serious Adverse Event (SAE) as follows:
  Serious Adverse Event (SAE)- an adverse event that:
  * results in death;
  * is life-threatening;
  * prolongs or results in hospitalization;
  * results in a persistent or significant disability;
  * causes a congenital anomaly or birth defect; or
  * is a medically significant event that jeopardizes the subject's health
Arm/Group | MoodGym Alone (Control) | Parenting Program + MoodGym (Intervention)
All-Cause Mortality (participants affected / at risk) | 0/37 | 0/38
Serious Adverse Events (participants affected / at risk) | 2/37 | 2/37
Other Adverse Events (participants affected / at risk) | 7/37 | 8/38
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MoodGym Alone (Control) (N=37) | Parenting Program + MoodGym (Intervention) (N=37)
Hospitalization-Breach of Confidentiality (Psychiatric disorders) | 2 (2) | 0 (0) — A breach of confidentiality occurred when a participant disclosed that they were hospitalized during the study (unrelated to study activities). Study personnel broke confidentiality and contacted social workers at the participant's child's clinic.
Hospitalization (Psychiatric disorders) | 0 (0) | 2 (2) — A participant disclosed that they were hospitalized during the study (unrelated to study activities). Participants consented to contact between the study team and the participant's child's doctor. The study team followed up and provided resources.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MoodGym Alone (Control) (N=37) | Parenting Program + MoodGym (Intervention) (N=38)
Protocol Deviation- Incorrect Version of Informed Consent (Psychiatric disorders) | 1 (1) | 2 (2) — A minor protocol deviation occurred and an older version of the informed consent was used. This version didn't include the section on arranged transportation. Participants were verbally informed during their visit about the transportation options.
Protocol Deviation- Unstamped Version of Informed Consent (Psychiatric disorders) | 6 (6) | 6 (6) — A minor protocol deviation occurred and a version of the informed consent was used that was not stamped by the IRB. The content of the unstamped ICF was identical to the IRB stamped version, the physical forms were just missing the IRB approval stamp

LIMITATIONS AND CAVEATS:
First, the study occurred in a single urban geographic area with a predominantly African-American population. Second, the study occurred during the height of the COVID-19 Pandemic. Third, engagement with the PWD Program was lower than expected.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-12-02): https://cdn.clinicaltrials.gov/large-docs/32/NCT04045132/Prot_SAP_000.pdf
  • Informed Consent Form (2020-12-08): https://cdn.clinicaltrials.gov/large-docs/32/NCT04045132/ICF_001.pdf